CLINICAL TRIAL: NCT03438864
Title: Acute Effects of Interferential Current on Edema, Pain and Muscle Strength in Patients With Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Funda Atamaz Calis, Professor in Department of Physical Medicine and Rehabilitation, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IF-Edema
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Radius Fractures; Edema; Pain
Keywords: Radius fracture, Interferential current, edema, pain
MeSH Terms: conditions — Radius Fractures; Edema; Pain | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 Hz (Experimental): Interferential current, entry frequency 4000 Hz and 4010 Hz, beat frequency 10 Hz, amplitude was individualized and increased until patients felt a comfortable tickling sensation.
  Interventions: Device: Electrotherapy, interferential current
- 100 Hz (Experimental): Interferential current, entry frequency 4000 Hz and 4100 Hz, beat frequency 100 Hz, amplitude was individualized and increased until patients felt a comfortable tickling sensation.
  Interventions: Device: Electrotherapy, interferential current
- Placebo-Sham Control (Sham Comparator): No current except for first 5 seconds, device open but does not appy electrotherapy.
  Interventions: Other: Control

INTERVENTIONS:
Device: Electrotherapy, interferential current — Interferential current, entry frequencies and beat frequencies were set differently in 2 groups, amplitude was individualized and increased until patients felt a comfortable tickling sensation.
  Arms: 10 Hz; 100 Hz
Other: Control — No current except for first 5 seconds, device open but does not appy electrotherapy.
  Arms: Placebo-Sham Control

SUMMARY:
Interferential current is a form of electrotherapy that is obtained by placing two different plates that produce medium frequency waveform current, resulting in a low frequency interferential waveform in deeper tissues. It was shown interferential current electrotherapy is beneficial for reduction of traumatic edema in tissues and pain control.

Patients with conservatively managed distal radius fractures were recruited after casts are shed, and were treated with one session(30 minutes) of different protocols of interferential current electrotherapy. Before and after therapy, they were evaluated with volumetry, hand grip strength and visual analogue scale for pain.

ELIGIBILITY:
Inclusion Criteria:

* Conservatively managed distal radius fractures

Exclusion Criteria:

* Secondary conditions associated with edema(renal failure, congestive heart failure etc)
* Complex regional pain syndrome
* Compartment syndrome
* Contraindications for electrotherapy(cardiac pacemaker, thrombosis, pregnancy etc)
* Mental state unfit for electrotherapy
* Having treated with electrotherapy before

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-01-07 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Volumetry | 30 minutes
  Patients were asked to dip their hands slowly into a special bucket full of water with volume markings until their middle finger touched to the bottom of the bucket. The spilled amount of water were measured as milliliters.
Visual Analogue Scale | 30 minutes
  Patients were asked to express their discomfort level from pain in a scale ranging from 1 to 10(with the help of a 10 cm line), and point they showed were measured as millimeters.
Hand Grip Strength | 30 minutes
  Patients were asked to use a hydraulic hand dynamometer for hand grip strength in a position of 10 to 30 degrees of wrist extension, and results were registered as kilograms.

IPD SHARING:
Plan to Share IPD: Undecided